CLINICAL TRIAL: NCT03408639
Title: A Phase III, Randomized, Two Armed, Parallel, Double Blind (Patient and Assessor Blinded), Active Controlled Non Inferiority Clinical Trial to Determine the Non Inferior Therapeutic Efficacy and Safety Between CinnaPoietin® (Beta Erythropoietin) and Eprex® (Epoetin Alpha) on the Treatment of Anemia in ESRD Hemodialysis Patients
Brief Title: Comparing Efficacy and Safety of CinnaGen Beta Erythropoietin (CinnaPoietin®) Versus Eprex® on the Treatment of Anemia in ESRD Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERY.CIN.MA.94; IRCT201601156135N6 (Other: Food And Drug Administration of The Islamic Republic of Iran)
Record Dates: First submitted 2017-12-12; First posted 2018-01-24 (Actual); Results first posted 2019-11-06 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Anemia in End-Stage Renal Disease
Keywords: End-Stage Renal Disease, Anemia, Erythropoietin, Hemoglobin
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Epoetin Alfa; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CinnaPoietin® (Experimental): The starting dose of Erythropoietin is 60 (50-100) IU/kg body weight/week for naïve patients. Administration dose for patients who are treated with erythropoietin is similar dose of previously administered amount (IV or SC without any change). After then, dose adjustment will be done based on patients' response.
  In addition to main intervention, Nephrovit tablet/day and vitamine B12 100 mcg/month will be prescribed for patients.
  Interventions: Drug: CinnaPoietin®; Drug: Nephrovit; Drug: Vitamin B12 Injection
- Eprex® (Active Comparator): The starting dose of Erythropoietin is 60 (50-100) IU/kg body weight/week for naïve patients. Administration dose for patients who are treated with erythropoietin is similar dose of previously administered amount (IV or SC without any change). After then, dose adjustment will be done based on patients' response. In addition to main intervention, Nephrovit tablet/day and vitamine B12 100 mcg/month will be prescribed for patients.
  Interventions: Drug: Eprex®; Drug: Nephrovit; Drug: Vitamin B12 Injection

INTERVENTIONS:
Drug: CinnaPoietin® — The starting dose of Erythropoietin is 60 (50-100) IU/kg body weight/week for naïve patients. Administration dose for patients who are treated with erythropoietin is similar dose of previously administered amount (IV or SC without any change). After then, dose adjustment will be done based on patients' response.
  Other Names: Beta erythropoietin
  Arms: CinnaPoietin®
Drug: Eprex® — The starting dose of Erythropoietin is 60 (50-100) IU/kg body weight/week for naïve patients. Administration dose for patients who are treated with erythropoietin is similar dose of previously administered amount (IV or SC without any change). After then, dose adjustment will be done based on patients' response.
  Other Names: Epoetin alpha
  Arms: Eprex®
Drug: Nephrovit — Nephrovit tablet is daily administered to all the patients.
Drug: Vitamin B12 Injection — Vitamin B12 is monthly injected to all the patients.

SUMMARY:
This Phase III, randomized, two-armed, parallel, double-blind, active-controlled clinical trial is designed to compare efficacy and safety of CinnaPoietin® (Beta erythropoietin) and Eprex® (epoetin alpha) on the treatment of anemia in 156 End-Stage Renal Disease hemodialysis patients. 156 patients have been planned to randomize and assign to receive CinnaPoietin® or Eprex® for a 26-week period. Administration dose for patients who are treated with erythropoietin is the similar dose of the previously administered amount (IV or SC without any change). After then, dose adjustment will be made based on patients' response. The primary objective of this study is to compare the efficacy of CinnaPoietin® with Eprex®. The secondary objectives of this study are further comparison and evaluation of efficacy along with safety between CinnaPoietin® and Eprex®.

DETAILED DESCRIPTION:
This study is a phase III, randomized, two-armed, parallel, double-blind (patient and assessor blinded), active-controlled noninferiority clinical trial to determine the non-inferior therapeutic efficacy and safety between CinnaPoietin® (Beta erythropoietin) and Eprex® (epoetin alpha) on the treatment of anemia in ESRD patient under hemodialysis. After signing the written informed consents, 156 patients have been planned to randomize and assign to receive CinnaPoietin® or Eprex® for a 26-weeks period. Administration dose for patients who are treated with erythropoietin is the similar dose of the previously administered amount (IV or SC without any change). After then, dose adjustment will be made based on patients' response. In addition to main intervention, Nephrovit tablet/day and B12 100 mcg/month were prescribed for patients. The primary objective of this study is to compare the efficacy of CinnaPoietin® with Eprex®. The secondary objectives of this study are further comparison and evaluation of efficacy and safety.

The clinical trial will be conducted according to the GCP considerations. A comprehensive validation check program is used to verify the data, and discrepancy reports are generated accordingly for resolution by the investigator.

In order to ensure the use of standard and unified procedure of each test, monitoring of each site and laboratory site are going to be applied by sponsor monitoring team and CRO as external monitoring team.

The same prefilled syringe is used for CinnaPoietin® to be sure that there is no difference between CinnaPoietin® and Eprex® as brand drug. The drugs will be relabeled, and the same label is used for both prefilled syringe. So neither investigators nor subjects are able to notice any differences between them and are blind to the assignment.

Determination of sample size 156 patients will be equally (1:1) divided into intervention arms (78 in each group considering drop out) for achieving 80% power in order to determine non-inferiority using a one-sided, independent sample t-test. The margin of non-inferiority is -1.00.

The true difference between the means is assumed to be -0.500. The significance level (alpha) of the test is 0.05. The data are drawn from populations with standard deviations of 1.200 and 1.200.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70
* ESRD patients who are on hemodialysis for ≥3 months.
* Hb level 8- 11.5 g/dl
* Patients are on adequate hemodialysis: the minimally adequate dose of hemodialysis given 3 times per week should be a spKt/V (single-pool delivered Kt/V; clearance of urea x dialysis time/volume of distribution) of 1.2 per dialysis. For treatment periods of less than 5 hours, an alternative minimum dose is a urea reduction rate (URR) of 65%. All types of hemodialysis systems and hemodiafiltration, including high-flux membranes are allowed as long as there is no plan to change the patient's regimen during the study.
* Sufficient iron stores, defined as serum ferritin ≥ 200 ng/ml and transferrin saturation ≥20%. (Patients not meeting these criteria may receive iron supplementation therapy during the Screening and stabilization period to appropriately correct their iron store deficiency to meet the criterion required for randomization);
* Ability to comply with study medication use, study visits, and study procedures as judged by the investigator;
* Females of childbearing potential agree to use an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or IUD) for the duration of the study.
* Qualified and willing to sign the informed consent form with the commitment of complying with all the scheduled visits, and study procedures as judged by the investigator;
* In any circumstances that potential participants are not able to give consent, it may be given by responsible parents or guardian.

Exclusion Criteria:

* Uncontrolled hypertension (defined as pre-dialysis diastolic blood pressure ≥ 100 mmHg or systolic blood pressure ≥180 mmHg);
* Anemia secondary to other causes different to the CKD (e.g. multiple myeloma, aplastic anemia, leukemia;….)
* Decompensated liver failure;
* Clinical evidence of concurrent uncontrolled hyperparathyroidism (defined as serum parathyroid hormone (iPTH) > 800 pg/ml);
* Heart failure [New York Heart Association (NYHA) class III and IV];
* Unstable angina pectoris, active cardiac disease, stroke and/or cardiac infarction within the last 6 months;
* History of or active blood coagulation disorders including DVT, PTE, native access Thrombosis during last 6 months.
* Thrombocytosis (platelet count > 500,000/µl);
* Thrombocytopenia (platelet count < 100,000/µl);
* White blood cell count < 3,000/µl);
* White blood cell count >15,000/µl)
* Recent Bleeding (acute or chronic bleeding within three months prior to screening);
* Suspicion of or confirmed occult bleeding (increased reticulocyte count);
* Clinical evidence of concurrent systemic infection, or inflammatory disease (e.g; diabetic foot, bed sore, access infection, CRP> 30 mg/l,…)
* Currently receiving treatment for epilepsy;
* Major surgery within 3 months prior to randomization and during the conduct of the trial (except vascular access surgery);
* Concomitant immunosuppressive therapy; patients on a short course of steroids (up to 7 days), topical or intranasal steroids are allowed in the study;
* History of any malignant disease within the last 5 years (except excised non-melanoma skin cancer);
* Women who are pregnant or breastfeeding;
* Known history of severe drug-related allergies;
* Known history of drug related allergy to Erythropoietin or one of the ingredients of the test or the reference products or hypersensitivity to mammalian-derived products;
* Transplant received within one year prior to the start of the study;
* Simultaneous participation in another clinical study or having received an Investigational Medicinal Product within three months before randomization in this study.
* Psychiatric, addictive (drugs or alcohol) or any other disorder that compromises the ability to give an informed consent;
* Any red blood cell transfusion during the last 3 months (measured at the time of eligibility verification);
* Primary hematological disorder (e.g. myelodysplastic syndrome, myeloma, sickle cell anemia, hematological malignancy, multiple myeloma hemolytic anemia);
* known resistance to the rHuEPO defined by a requirement > 450 IU/kg/week by IV or 300 IU/kg/week by SC, equivalent to approximately 20.000 IU/week SC and in absence of iron deficiency;
* who have suffered an event of active bleeding in the 30 days prior to the beginning of the study;
* Morbid obesity, defined by a Body Mass Index (BMI) > 37 kg/m2 in women and > 40 kg/m2 in men.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Iran (8):
  - Javad-al-Aemeh clinic, Kerman
  - SHAFA Hospital, Kerman
  - Haj Ebrahimi dialysis center, Shiraz
  - Ghiasi hospital, Tehran
  - Hashemi Nezhad Hospital, Tehran
  - Imam Hussein Hospital, Tehran
  - Madar dialysis center, Tehran
  - Milad Hospital, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astor BC, Muntner P, Levin A, Eustace JA, Coresh J. Association of kidney function with anemia: the Third National Health and Nutrition Examination Survey (1988-1994). Arch Intern Med. 2002 Jun 24;162(12):1401-8. doi: 10.1001/archinte.162.12.1401. PMID 12076240
- [Background] McLean E, Cogswell M, Egli I, Wojdyla D, de Benoist B. Worldwide prevalence of anaemia, WHO Vitamin and Mineral Nutrition Information System, 1993-2005. Public Health Nutr. 2009 Apr;12(4):444-54. doi: 10.1017/S1368980008002401. Epub 2008 May 23. PMID 18498676
- [Background] Brittin GM, Brecher G, Johnson CA, Elashoff RM. Stability of blood in commonly used anticoagulants. Use of refrigerated blood for quality control of the Coulter Counter Model S. Am J Clin Pathol. 1969 Dec;52(6):690-4. doi: 10.1093/ajcp/52.6.690. No abstract available. PMID 4982112
- [Background] Locatelli F, Aljama P, Barany P, Canaud B, Carrera F, Eckardt KU, Horl WH, Macdougal IC, Macleod A, Wiecek A, Cameron S; European Best Practice Guidelines Working Group. Revised European best practice guidelines for the management of anaemia in patients with chronic renal failure. Nephrol Dial Transplant. 2004 May;19 Suppl 2:ii1-47. doi: 10.1093/ndt/gfh1032. No abstract available. PMID 15206425
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Fehr T, Ammann P, Garzoni D, Korte W, Fierz W, Rickli H, Wuthrich RP. Interpretation of erythropoietin levels in patients with various degrees of renal insufficiency and anemia. Kidney Int. 2004 Sep;66(3):1206-11. doi: 10.1111/j.1523-1755.2004.00880.x. PMID 15327419
- [Background] Ross RP, McCrea JB, Besarab A. Erythropoietin response to blood loss in hemodialysis patients in blunted but preserved. ASAIO J. 1994 Jul-Sep;40(3):M880-5. doi: 10.1097/00002480-199407000-00122. PMID 8555638
- [Background] Lipschitz DA, Cook JD, Finch CA. A clinical evaluation of serum ferritin as an index of iron stores. N Engl J Med. 1974 May 30;290(22):1213-6. doi: 10.1056/NEJM197405302902201. No abstract available. PMID 4825851
- [Background] Rambod M, Kovesdy CP, Kalantar-Zadeh K. Combined high serum ferritin and low iron saturation in hemodialysis patients: the role of inflammation. Clin J Am Soc Nephrol. 2008 Nov;3(6):1691-701. doi: 10.2215/CJN.01070308. Epub 2008 Oct 15. PMID 18922994
- [Background] Fernandez-Rodriguez AM, Guindeo-Casasus MC, Molero-Labarta T, Dominguez-Cabrera C, Hortal-Casc n L, Perez-Borges P, Vega-Diaz N, Saavedra-Santana P, Palop-Cubillo L. Diagnosis of iron deficiency in chronic renal failure. Am J Kidney Dis. 1999 Sep;34(3):508-13. doi: 10.1016/s0272-6386(99)70079-x. PMID 10469862
- [Background] Kalantar-Zadeh K, Hoffken B, Wunsch H, Fink H, Kleiner M, Luft FC. Diagnosis of iron deficiency anemia in renal failure patients during the post-erythropoietin era. Am J Kidney Dis. 1995 Aug;26(2):292-9. doi: 10.1016/0272-6386(95)90649-5. PMID 7645533
- [Background] Aljama P, Ward MK, Pierides AM, Eastham EJ, Ellis HA, Feest TG, Conceicao S, Kerr DN. Serum ferritin concentration: a reliable guide to iron overload in uremic and hemodialyzed patients. Clin Nephrol. 1978 Sep;10(3):101-4. PMID 699405
- [Background] Barany P, Eriksson LC, Hultcrantz R, Pettersson E, Bergstrom J. Serum ferritin and tissue iron in anemic dialysis patients. Miner Electrolyte Metab. 1997;23(3-6):273-6. PMID 9387132
- [Background] Blumberg AB, Marti HR, Graber CG. Serum ferritin and bone marrow iron in patients undergoing continuous ambulatory peritoneal dialysis. JAMA. 1983 Dec 23-30;250(24):3317-9. PMID 6645029
- [Background] Hussein S, Prieto J, O'Shea M, Hoffbrand AV, Baillod RA, Moorhead JF. Serum ferritin assay and iron status in chronic renal failure and haemodialysis. Br Med J. 1975 Mar 8;1(5957):546-8. doi: 10.1136/bmj.1.5957.546. PMID 49205
- [Background] Mirahmadi KS, Paul WL, Winer RL, Dabir-Vaziri N, Byer B, Gorman JT, Rosen SM. Serum ferritin level. Determinant of iron requirement in hemodialysis patients. JAMA. 1977 Aug 15;238(7):601-3. doi: 10.1001/jama.238.7.601. PMID 577960
- [Background] Spinowitz BS, Kausz AT, Baptista J, Noble SD, Sothinathan R, Bernardo MV, Brenner L, Pereira BJ. Ferumoxytol for treating iron deficiency anemia in CKD. J Am Soc Nephrol. 2008 Aug;19(8):1599-605. doi: 10.1681/ASN.2007101156. Epub 2008 Jun 4. PMID 18525001
- [Background] Silverberg DS, Blum M, Agbaria Z, Deutsch V, Irony M, Schwartz D, Baruch R, Yachnin T, Steinbruch S, Iaina A. The effect of i.v. iron alone or in combination with low-dose erythropoietin in the rapid correction of anemia of chronic renal failure in the predialysis period. Clin Nephrol. 2001 Mar;55(3):212-9. PMID 11316241
- [Background] Stancu S, Barsan L, Stanciu A, Mircescu G. Can the response to iron therapy be predicted in anemic nondialysis patients with chronic kidney disease? Clin J Am Soc Nephrol. 2010 Mar;5(3):409-16. doi: 10.2215/CJN.04280609. Epub 2009 Dec 17. PMID 20019121
- [Background] Fishbane S, Frei GL, Maesaka J. Reduction in recombinant human erythropoietin doses by the use of chronic intravenous iron supplementation. Am J Kidney Dis. 1995 Jul;26(1):41-6. doi: 10.1016/0272-6386(95)90151-5. PMID 7611266
- [Background] Sunder-Plassmann G, Horl WH. Importance of iron supply for erythropoietin therapy. Nephrol Dial Transplant. 1995 Nov;10(11):2070-6. PMID 8643170
- [Background] Macdougall IC, Tucker B, Thompson J, Tomson CR, Baker LR, Raine AE. A randomized controlled study of iron supplementation in patients treated with erythropoietin. Kidney Int. 1996 Nov;50(5):1694-9. doi: 10.1038/ki.1996.487. PMID 8914038
- [Background] Chang CH, Chang CC, Chiang SS. Reduction in erythropoietin doses by the use of chronic intravenous iron supplementation in iron-replete hemodialysis patients. Clin Nephrol. 2002 Feb;57(2):136-41. doi: 10.5414/cnp57136. PMID 11863124
- [Background] DeVita MV, Frumkin D, Mittal S, Kamran A, Fishbane S, Michelis MF. Targeting higher ferritin concentrations with intravenous iron dextran lowers erythropoietin requirement in hemodialysis patients. Clin Nephrol. 2003 Nov;60(5):335-40. doi: 10.5414/cnp60335. PMID 14640239
- [Background] Rozen-Zvi B, Gafter-Gvili A, Paul M, Leibovici L, Shpilberg O, Gafter U. Intravenous versus oral iron supplementation for the treatment of anemia in CKD: systematic review and meta-analysis. Am J Kidney Dis. 2008 Nov;52(5):897-906. doi: 10.1053/j.ajkd.2008.05.033. Epub 2008 Oct 8. PMID 18845368
- [Background] Senger JM, Weiss RJ. Hematologic and erythropoietin responses to iron dextran in the hemodialysis environment. ANNA J. 1996 Jun;23(3):319-23; discussion 324-5. PMID 8716991
- [Background] Navarro JF, Teruel JL, Liano F, Marcen R, Ortuno J. Effectiveness of intravenous administration of Fe-gluconate-Na complex to maintain adequate body iron stores in hemodialysis patients. Am J Nephrol. 1996;16(4):268-72. doi: 10.1159/000169008. PMID 8739277
- [Background] Tessitore N, Solero GP, Lippi G, Bassi A, Faccini GB, Bedogna V, Gammaro L, Brocco G, Restivo G, Bernich P, Lupo A, Maschio G. The role of iron status markers in predicting response to intravenous iron in haemodialysis patients on maintenance erythropoietin. Nephrol Dial Transplant. 2001 Jul;16(7):1416-23. doi: 10.1093/ndt/16.7.1416. PMID 11427634
- [Background] Van Wyck DB, Roppolo M, Martinez CO, Mazey RM, McMurray S; United States Iron Sucrose (Venofer) Clinical Trials Group. A randomized, controlled trial comparing IV iron sucrose to oral iron in anemic patients with nondialysis-dependent CKD. Kidney Int. 2005 Dec;68(6):2846-56. doi: 10.1111/j.1523-1755.2005.00758.x. PMID 16316362
- [Background] Allegra V, Mengozzi G, Vasile A. Iron deficiency in maintenance hemodialysis patients: assessment of diagnosis criteria and of three different iron treatments. Nephron. 1991;57(2):175-82. doi: 10.1159/000186246. PMID 1902285
- [Background] Li H, Wang SX. Intravenous iron sucrose in Chinese hemodialysis patients with renal anemia. Blood Purif. 2008;26(2):151-6. doi: 10.1159/000113529. Epub 2008 Jan 22. PMID 18212498
- [Background] Palmer SC, Navaneethan SD, Craig JC, Johnson DW, Tonelli M, Garg AX, Pellegrini F, Ravani P, Jardine M, Perkovic V, Graziano G, McGee R, Nicolucci A, Tognoni G, Strippoli GF. Meta-analysis: erythropoiesis-stimulating agents in patients with chronic kidney disease. Ann Intern Med. 2010 Jul 6;153(1):23-33. doi: 10.7326/0003-4819-153-1-201007060-00252. Epub 2010 Jun 24. PMID 20439566
- [Background] Parfrey PS, Wish T. Quality of life in CKD patients treated with erythropoiesis-stimulating agents. Am J Kidney Dis. 2010 Mar;55(3):423-5. doi: 10.1053/j.ajkd.2009.12.014. No abstract available. PMID 20189050
- [Background] Gandra SR, Finkelstein FO, Bennett AV, Lewis EF, Brazg T, Martin ML. Impact of erythropoiesis-stimulating agents on energy and physical function in nondialysis CKD patients with anemia: a systematic review. Am J Kidney Dis. 2010 Mar;55(3):519-34. doi: 10.1053/j.ajkd.2009.09.019. Epub 2009 Dec 23. PMID 20031287
- [Background] Johansen KL, Finkelstein FO, Revicki DA, Gitlin M, Evans C, Mayne TJ. Systematic review and meta-analysis of exercise tolerance and physical functioning in dialysis patients treated with erythropoiesis-stimulating agents. Am J Kidney Dis. 2010 Mar;55(3):535-48. doi: 10.1053/j.ajkd.2009.12.018. Epub 2010 Feb 4. PMID 20133033
- [Background] Solomon SD, Uno H, Lewis EF, Eckardt KU, Lin J, Burdmann EA, de Zeeuw D, Ivanovich P, Levey AS, Parfrey P, Remuzzi G, Singh AK, Toto R, Huang F, Rossert J, McMurray JJ, Pfeffer MA; Trial to Reduce Cardiovascular Events with Aranesp Therapy (TREAT) Investigators. Erythropoietic response and outcomes in kidney disease and type 2 diabetes. N Engl J Med. 2010 Sep 16;363(12):1146-55. doi: 10.1056/NEJMoa1005109. PMID 20843249
- [Derived] Azmandian J, Abbasi MR, Pourfarziani V, Nasiri AA, Ossareh S, Ezzatzadegan Jahromi S, Sanadgol H, Amini S, Shahvaroughi Farahani A. Comparing Therapeutic Efficacy and Safety of Epoetin Beta and Epoetin Alfa in the Treatment of Anemia in End-Stage Renal Disease Hemodialysis Patients. Am J Nephrol. 2018;48(4):251-259. doi: 10.1159/000493097. Epub 2018 Sep 25. PMID 30253403

RESULTS

PARTICIPANT FLOW:
Groups:
- CinnaPoietin®: The starting dose of Erythropoietin is 60 (50-100) IU/kg body weight/week for naïve patients. Administration dose for patients who are treated with erythropoietin is similar dose of previously administered amount (IV or SC without any change). After then, dose adjustment will be done based on patients' response.
  In addition to main intervention, Nephrovit tablet/day and vitamine B12 100 mcg/month will be prescribed for patients.
  CinnaPoietin®: The starting dose of Erythropoietin is 60 (50-100) IU/kg body weight/week for naïve patients. Administration dose for patients who are treated with erythropoietin is similar dose of previously administered amount (IV or SC without any change). After then, dose adjustment will be done based on patients' response.
  Nephrovit: Nephrovit tablet is daily administered to all the patients.
  Vitamin B12 Injection: Vitamin B12 is monthly injected to all the patients.
Period: Overall Study
Arm/Group | CinnaPoietin® | Eprex®
Started | 78 | 78
Completed | 67 | 56
Not Completed | 11 | 22
Not completed — Death | 5 | 5
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Physician Decision | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CinnaPoietin® | Eprex® | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 69 | 129
  >=65 years | 18 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.02 (11.38) | 50.01 (12.72) | 52.53 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 45 | 45 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 78 | 78 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Iran | 78 | 78 | 156
Hemoglobin concentration [Mean (Standard Deviation); unit: g/dL] | 10.41 (0.89) | 10.64 (0.82) | 10.53 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: Mean Hb Change Level During the Last Four Weeks of Treatment
Description: The primary endpoints of this study is to assess mean Hb change level during the last four weeks of treatment.
Time Frame: Week 22 to week 26
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 61 | 38
g/dL | 0.4 (1.26) | 0.74 (1.39)

2. Primary Outcome: Mean Weekly Epoetin Dosage Per kg Body Weight During the Last Four Weeks of Treatment
Description: The mean weekly epoetin dosage per kg body weight during the last four weeks of treatment necessary to maintain the Hb level within 10-12 g/dl during the last four weeks of treatment is considered as the second primary endpoint.
Time Frame: Week 22 to week 26
Measure: Mean (Standard Deviation); unit: IU/Kg/week
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 46 | 19
IU/Kg/week | 117.02 (54.5) | 110.01 (49.27)

3. Secondary Outcome: The Proportion of Patients With Any Permanent or Transient Dose Change
Description: The proportion of patients with any permanent or transient dose change during 26 weeks.
Time Frame: 26 weeks
Measure: Number; unit: proportion of patients
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 72 | 66
proportion of patients | 0.9 | 0.95

4. Secondary Outcome: The Proportion of Patients With Any Hb Measurement Outside the Target Range (10-12 g/dl)
Description: The proportion of patients with any Hb measurement outside the target range (10-12 g/dl) during 26 weeks.
Time Frame: 26 weeks
Measure: Number; unit: proportion of patients
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 74 | 73
proportion of patients | 0.92 | 1

5. Secondary Outcome: The Proportion of Patients Needed Blood Transfusions
Description: The proportion of patients needed blood transfusions during 26 weeks.
Time Frame: 26 weeks
Measure: Number; unit: proportion of patients
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 78 | 78
proportion of patients | 0.04 | 0.04

6. Secondary Outcome: The Proportion of Patients With Treatment Success
Description: Treatment success is considered as Hb concentration equal to or more than 11.0 g/dl and two consecutive weeks without any blood transfusion within the preceding three months
Time Frame: Week 12 to week 26
Measure: Number; unit: proportion of patients
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 54 | 25
proportion of patients | 0.41 | 0.44

7. Secondary Outcome: The Proportion of Patients With Maintenance Success
Description: Maintenance success is considered as maintenance success is considered as maintenance of mean Hb concentration of 11.0 ± 1.0 g/dl for at least four consecutive weeks
Time Frame: 26 weeks
Measure: Number; unit: proportion of patients
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 68 | 56
proportion of patients | 0.71 | 0.43

8. Secondary Outcome: The Percentage of Patients With Hb Measurements More Than 10.0 g/dl
Description: The percentage of patients with Hb measurements more than 10.0 g/dl from week 22 to week 26.
Time Frame: Week 22 to week 26
Measure: Count of Participants; unit: Participants
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 68 | 56
Participants | 55 | 48

9. Secondary Outcome: The Percentage of Patients With Hematocrit Measurements More Than 30%
Description: The percentage of patients with hematocrit measurements more than 30% from week 22 to week 26.
Time Frame: Week 22 to week 26
Measure: Number; unit: percentage of patients
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 68 | 56
percentage of patients | 86.76 | 92.86

10. Secondary Outcome: The Incidence of Hb Levels Above 13 g/dl
Description: The first safety endpoint is the proportion of patients with at least one Hb measurement above 13 g/dL.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 70 | 59
Participants | 31 | 42

11. Secondary Outcome: The Proportion of Patients With an Increase in Hb Concentration of > 1.0 g/dl for Four Consecutive Weeks
Description: The proportion of patients with an increase in Hb concentration of > 1.0 g/dl for four consecutive weeks during 26 weeks.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 72 | 65
Participants | 44 | 41

12. Secondary Outcome: The Incidence of Adverse Events
Description: The incidence of adverse events during 26 weeks.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CinnaPoietin® | Eprex®
Number analyzed (Participants) | 78 | 78
Participants | 23 | 18

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | CinnaPoietin® | Eprex®
All-Cause Mortality (participants affected / at risk) | 5/78 | 5/78
Serious Adverse Events (participants affected / at risk) | 14/78 | 7/78
Other Adverse Events (participants affected / at risk) | 11/78 | 12/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CinnaPoietin® (N=78) | Eprex® (N=78)
Palpitation, Cardiac Function Impairment, Cardiac Infraction, Chest Pain, Tachycardia) (Cardiac disorders) | 2 | 3
Inflation on Ankle (Renal and urinary disorders) | 1 | 0
(Skin reaction, Catheter defect, Disability catheter, Filter clots, pain in injection site, skin rea (General disorders) | 4 | 0
Gallstones (Hepatobiliary disorders) | 1 | 0
(Pneumonia, Infection of right hand Lower than the fistula) (Infections and infestations) | 2 | 0
(CO toxicity, transplantation complication) (Injury, poisoning and procedural complications) | 0 | 2
(tearing of tendon in both knees, back pain, Musculoskeletal-Bone pain, knee tenderness due to joint (Musculoskeletal and connective tissue disorders) | 2 | 1
(Respiratory disorder, chest pain and dyspenea, dyspnea) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
echymosis due to recent car accident, itching) (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac pacemaker AND Valve Replacement, orthopedic surgery) (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CinnaPoietin® (N=78) | Eprex® (N=78)
(Eosinophilia, Thrombocytopenia) (Blood and lymphatic system disorders) | 0 | 1
(Palpitation, Cardiac Function Impairment, Cardiac Infraction, Chest Pain, Tachycardia) (Cardiac disorders) | 1 | 3
(Skin reaction, Catheter defect, Disability catheter, Filter clots, pain in injection site, skin rea (General disorders) | 3 | 1
(Pneumonia, Infection of right hand Lower than the fistula) (Infections and infestations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
(tearing of tendon in both knees, back pain, Musculoskeletal-Bone pain, knee tenderness due to joint (Musculoskeletal and connective tissue disorders) | 0 | 1
(numbness in the wrist, dizziness) (Nervous system disorders) | 1 | 1
Decreased libido (Psychiatric disorders) | 1 | 0
vaginal discharge (Reproductive system and breast disorders) | 0 | 1
(Respiratory disorder, chest pain and dyspenea, dyspnea) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
(itching, echymosis due to recent car accident, itching) (Skin and subcutaneous tissue disorders) | 0 | 2
(Installing Cardiac pacemaker AND Valve Replacement, orthopedic surgery) (Surgical and medical procedures) | 0 | 1
(blood clotting, Bleeding catheter, Hemorrage, Vascular disorders) (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator (PI) may publish results provided a copy of the written publication is received by the sponsor at least 30 days in advance for review and comment. If the parties disagree, PI agrees to meet with the sponsor before submission to resolve any disagreement. It is also agreed that publishing any reports from data is under the condition of the subject's consent. Any reports are highly confidential, and the PI does not have the permission to reveal them without the sponsor's agreement.

DOCUMENTS (2):
  • Study Protocol (2015-08-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03408639/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT03408639/SAP_001.pdf